CLINICAL TRIAL: NCT04516148
Title: A Randomized, Controlled Trial of the Effectiveness of Perioperative Antibiotics for Reduction of Burn Wound Bacterial Concentration Following Grafting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017-186
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Burn; Surgery; Infection Wound
Keywords: microbiome; perioperative; antibiotics; autograft; xenograft
MeSH Terms: conditions — Burns; Wound Infection | interventions — Cefazolin; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Antibiotics (Experimental): Patients randomized to the treatment arm of the study will have orders placed by a physician on the clinical team, with preparation and delivery of the antibiotics dose by the pharmacy following standard procedures. Antibiotic administration will occur after induction of anesthesia, with delivery by the Anesthesia staff no more than one hour prior to incision. Those with known allergy to beta-lactams will receive clindamycin instead of cefazolin.
  Interventions: Drug: Cefazolin; Drug: Clindamycin
- Standard of Care (No Intervention): Patients randomized to the standard of care arm of the study will receive no perioperative antibiotic administration and will proceed with routine pre-operative care.

INTERVENTIONS:
Drug: Cefazolin — Dosing per hospital policy
  Arms: Antibiotics
Drug: Clindamycin — Dosing per hospital policy
  Arms: Antibiotics

SUMMARY:
The purpose of this study if to evaluate the effectiveness of prophylactic antibiotics given during surgery in reducing the concentration of bacteria in a burn wound after surgery.

DETAILED DESCRIPTION:
This is a single-blind, randomized, controlled study to assess the effectiveness and safety of prophylactic perioperative administration of antibiotics for the reduction of bacterial concentration in burn wounds. Subjects who meet enrollment criteria will be randomized in a 1:1 ratio to receive either perioperative prophylaxis with intravenous antibiotics or institutional standard of care, consisting of no antibiotic therapy. This with be a single center study.

Following randomization, patients will receive their assigned treatment (antibiotics or standard of care) after induction of anesthesia, no more than one hour prior to incision.

Patients weighing 120 kg or less will receive 2 grams of intravenous cefazolin, with those weighing > 120 kg receiving 3 grams intravenous cefazolin. Re-dosing will occur every 4 hours that the patient remains in the operating room.

For patients with a documented beta-lactam allergy, Clindamycin 900 mg will be given intravenously with re-dosing every 6 hours that the patient remains in the operating room. Patients with allergies to both agents will be excluded from the study.

Biological samples will be obtained at three primary time-points: intraoperatively, at the time of the initial postoperative dressing take-down (within six hours), and at the time of a single follow up visit (10-28 days postoperatively).

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18 years old at the time of consent
2. Burn wound sustained less than 48 hours prior to the time of presentation to MedStar Washington Hospital Center
3. Burn wounds solely due to a thermal mechanism
4. Total body surface area burned ≤ 10%
5. Anticipated to require a single grafting procedure
6. Able to provide informed consent to participate

Exclusion Criteria:

1. Positive pregnancy test in females of child bearing age
2. Antibiotic administration within 30 days prior to admission
3. Known / documented beta lactam allergy and clindamycin allergy
4. Presence of burn wound cellulitis or infection pre-operatively
5. Intraoperative discovery of infection
6. Incarceration
7. Presence of factors that may affect wound healing, per clinician judgment, such as chronic malnutrition and immunocompromised state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
burn wound bacterial concentration | 1-3 days from surgery
  The primary effectiveness endpoint is a statistically significant reduction in the burn wound bacterial concentration in wounds where patients received antibiotics. Samples (tissue swabs and punch biopsies) obtained intraoperatively following wound bed preparation will be compared to samples (tissue swabs and punch biopsies) obtained from the wound within six hours of initial postoperative dressing take-down.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States